CLINICAL TRIAL: NCT03681288
Title: Mindful Self Compassion for Combat Deployed Veterans With Moral Injury and Co-occurring PTSD-SUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Providence VA Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2893-P; 1I21RX002893-01A1 (NIH)
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Results first posted 2024-06-21 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-02

CONDITIONS: Substance Use Disorder; Post-traumatic Stress Disorder; Moral Injury
Keywords: PTSD; substance use disorder; moral injury; self-compassion; mindfulness; Veterans
MeSH Terms: conditions — Substance-Related Disorders; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Mindful Self-Compassion (Experimental): Mindful Self-Compassion Intervention
  Interventions: Behavioral: Mindful Self-Compassion

INTERVENTIONS:
Behavioral: Mindful Self-Compassion — Mindful Self-Compassion Intervention

SUMMARY:
Veterans with co-occurring Posttraumatic Stress Disorder and Substance Use Disorder (PTSD-SUD) experience more severe symptomatology and poorer response to existing treatments than Veterans with either disorder alone. Guilt is a common posttraumatic reaction and has been implicated as a risk factor for the development and maintenance of PTSD and substance use. Combat Veterans often report experiencing moral injury defined as perpetrating, failing to prevent, or witnessing acts that violate the values they live by in their civilian lives, which can lead to feelings of guilt and shame. Accordingly, reduction in guilt and increase in self-compassion may lead to improved quality of life for Veterans. This project will conduct a pilot study to evaluate changes in self-compassion, guilt, and PTSD-SUD symptom severity in a sample of Veterans after receiving 8 sessions of Mindful Self Compassion treatment (via a telehealth modality during COVID-19 pandemic). Findings will have significant impact on effective treatment options and lead to improvements in Veterans' quality of life and posttraumatic symptoms.

DETAILED DESCRIPTION:
PTSD-SUD is particularly common following combat exposure, affecting a rapidly increasing number of U.S. military Veterans. The co-occurrence of these disorders presents added challenges to the VA treatment delivery system, presently in need of effective integrated treatments. Veterans with PTSD-SUD experience more severe symptomatology, increased risk of suicidality, poorer quality of life, and poorer response to existing treatments than Veterans with either disorder alone. Furthermore, PTSD-SUD prevents Veterans from reintegrating into society and is associated with occupational and social dysfunction. These findings underscore the need to effectively and efficiently address comorbidity and the complex array of problems with which Veterans present to treatment.

One approach is to develop interventions that target mechanisms thought to underlie multiple highly prevalent disorders, such as guilt related to traumatic experiences. Combat Veterans often report experiencing moral injury defined as perpetrating, failing to prevent, or witnessing acts that violate the values they live by in their civilian lives. Veterans who negatively appraise their actions or inaction during combat may experience guilt, a common posttraumatic reaction. Moral injury suggests the inability to contextualize or justify actions and the unsuccessful accommodation of those morally challenging experiences into pre-existing moral schemas, resulting in guilt and shame. Posttraumatic guilt has been implicated as a risk factor for the development and maintenance of several forms of psychopathology including PTSD, SUD, depression, and suicidality. However, to date, treatments for posttraumatic psychological health issues have been primarily disorder specific, with a focus largely on symptom reduction. Therefore, greater understanding of modifiable factors that influence functional impairment and PTSD-SUD is needed to enhance treatment efforts.

Mindful Self Compassion (MSC) combines the skills of mindfulness and self-compassion, providing self-soothing skills to respond to difficult thoughts and feelings (including guilt) via meditation. Self-compassion (SC) emphasizes kindness towards one's self, a feeling of connectedness with others, and mindful awareness of distressing experiences. Furthermore, because SC is negatively associated with self-criticism, rumination, thought suppression, anxiety, and depression, and positively associated with healthy psychological functioning, it is well suited to addressing posttraumatic psychopathology, shame, and guilt.

This proposal will begin to address a gap in the field's knowledge about MSC, and its role in the treatment of co-occurring disorders in Veterans with moral injury. The investigators will evaluate changes in self-compassion, post-traumatic guilt, shame, PTSD and substance use symptom severity. In addition to symptom reduction, the investigators will focus on functional outcomes (e.g., quality of life, suicidality). Participants will complete assessments at baseline, post-treatment, and 1-month follow-up. This project will allow us to 1) determine the feasibility of recruitment, 2) determine the acceptability of MSC, 3) provide preliminary evidence of the effects of MSC, and 4) refine study procedures and make adaptations to MSC based upon experience gained in the pilot in preparation for a fully powered randomized control trial (RCT) to test the effectiveness of MSC.

ELIGIBILITY:
Inclusion Criteria:

* moral injury as captured by at least one "strongly agree" response on the Moral Injury Events Scale
* diagnosis of PTSD (within the last 30 days) confirmed by the Clinician Administered PTSD Scale (CAPS) with a total symptom score of 22 or more
* diagnosis of a substance use disorder confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual-5 (DSM-5) Section E (SCID-E) within the last year
* willing and able to provide informed consent
* not currently receiving trauma-focused treatment

Exclusion Criteria:

* individuals with an acute psychotic disorder or acute psychotic symptoms are not eligible if their symptoms are unstable and if they are not well connected with appropriate mental health services
* patients with a psychiatric hospitalization or suicide attempt within the past month will be excluded
* currently receiving trauma-focused treatment, e.g., (Prolonged Exposure (PE), Cognitive Processing Therapy (CPT), Cognitive Behavioral Therapy (CBT) for PTSD)

  * Patients currently enrolled in trauma-focused treatment may be enrolled when they have completed the treatment if they remain interested and continue to have PTSD
* individuals with life-threatening or unstable medical illness. Diagnoses of mild cognitive impairment (e.g. mTBI) and other anxiety and depressive disorders will not be excluded because of their high comorbidity with PTSD and SUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-07-08 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erica M. Eaton, PhD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared. The principal investigator will share de-identified datasets, statistics, and results collected from this proposal by depositing these data at the National Library of Medicine (NLM) PubMed Central website repository as this is a VA supported data repository. Additional documentation including metadata that will include information about the methodology and study procedures used to collect the data, details about code, and 'definition of variables will also be included.
  Both scientists and the public will benefit from sharing these data because data sharing incentivizes researchers to produce and ensure higher quality data for sharing with peers, the scientific community, and the public. Further, data sharing encourages collaboration among researchers to share resources to produce new findings and reduces redundancy of data production in scientific research, which saves investment dollars and time.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months post publication
Access Criteria: 6 months post publication

REFERENCES:
- [Derived] Eaton E, Capone C, Reese S, Shea MT, Serpa JG, Germer C. Mindful Self-Compassion for Veterans with Morally Injurious Experiences and Co-Occurring Posttraumatic Stress Disorder and Substance Use Disorder: A Feasibility Study. J Dual Diagn. 2025 Apr;21(2):87-98. doi: 10.1080/15504263.2025.2474953. Epub 2025 Apr 1. PMID 40168188

RESULTS

PARTICIPANT FLOW:
Recruitment Details: During a 18-month period, the investigators enrolled 34 patients who were referred or self-referred themselves to the Mindful Self-Compassion (MSC) program at the Providence VA Medical Center. 76.5% (n=26) of eligible participants who completed the baseline assessment enrolled in MSC by attending the first session.
Groups:
- Mindful Self-Compassion (MSC): Mindful Self-Compassion Intervention
Period: Overall Study
Arm/Group | Mindful Self-Compassion (MSC)
Started | 26
Completed | 18
Not Completed | 8

BASELINE CHARACTERISTICS:
Population: 34 veterans were recruited for an 8-week MSC group intervention and were eligible for participation in the MSC intervention. 76.5% (n=26) of eligible participants who completed the baseline assessment enrolled in MSC by attending the first session.
Arm/Group | Mindful Self-Compassion (MSC)
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.92 (15.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino: Hispanic or Latino | 0
  Hispanic or Latino: Not Hispanic or Latino | 26
  Hispanic or Latino: Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Education Level [Count of Participants; unit: Participants]
  High School Grad/GED | 6
  Some College/Technical School | 13
  College Graduate | 2
  Post-Graduate/Professional Degree | 5
Relationship Status [Count of Participants; unit: Participants]
  Single | 5
  Married or in a committed relationship (living together) | 15
  Separated | 1
  Divorced | 5
Clinician Administered PTSD Scale (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — Clinician Administered PTSD Scale for DSM-5 (CAPS-5; range 0-80; higher scores indicate worse PTSD) was administered to assess diagnostic criteria for PTSD . Participants must meet criteria on this measure, considered the "gold standard" for PTSD diagnosis, to be eligible for the study. Participants must also have a total score of 23 or greater, which constitutes at least a moderate (or clinically significant) level of symptom severity. The follow-up version will be used at post-treatment and at 1-month follow-up as a primary measure of outcome.
  units on a scale | 41.33 (8.98)
PTSD Checklist (PCL-5) [Mean (Standard Deviation); unit: units on a scale] — The PCL-5 is a 20-item self-report measure that assesses DSM-5 symptoms of PTSD and PTSD symptom severity on a 5-point scale. The self-report rating scale is 0-4 for each symptom, from "Not at all" to "Extremely." A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items. DSM-5 symptom cluster severity scores can be obtained by summing the scores for the items within a given cluster, i.e., cluster B (items 1-5), cluster C (items 6-7), cluster D (items 8-14), and cluster E (items 15-20). Higher scores indicate worse PTSD symptoms.
  units on a scale | 57.67 (17.01)
Trauma Related Guilt Inventory (TRGI) - Distress Subscale [Mean (Standard Deviation); unit: units on a scale] — The TRGI distress subscale is made up of 6 items (e.g., "I experience severe emotional distress when I think about what happened"). Respondents rate each statement using a 5-point Likert scale to indicate the degree to which they believe the statement is true about themselves (i.e., Extremely True=4, Very True=3, Somewhat True=2, Slightly True=1, or Never True=0). The items are summed and divided by 6 to create an average score raging from 0-4 with higher scores reflecting higher levels of distress.
  units on a scale | 3.05 (.93)
Trauma Related Guilt Inventory (TRGI) - Global Guilt Subscale [Mean (Standard Deviation); unit: units on a scale] — The TRGI global guilt subscale is made up of 4 items (e.g., "I experience intense guilt that relates to what happened"). Respondents rate each statement using a 5-point Likert scale to indicate the degree to which they believe the statement is true about themselves (i.e., Extremely True=4, Very True=3, Somewhat True=2, Slightly True=1, or Never True=0). Items are summed (with three of the items being reverse scored) and divided by 4 to create an average score (range 0-4). Higher scores reflect higher levels of global guilt.
  units on a scale | 1.83 (.61)
Trauma Related Guilt Inventory (TRGI) - Guilt Cognitions Subscale [Mean (Standard Deviation); unit: units on a scale] — The TRGI guilt cognitions subscale is 22 items (e.g., "What I did was unforgivable"). Respondents rate each statement using a 5-point Likert scale to indicate the degree to which they believe the statement is true about themselves (i.e., Extremely True=4, Very True=3, Somewhat True=2, Slightly True=1, or Never True=0). Items are summed (with four of the items being reverse scored) and divided by 22 to create an average score (range 0-4). Higher scores reflect increased severity of guilt cognitions.
  units on a scale | 1.58 (.84)
Trauma Related Shame Inventory (TRSI) [Mean (Standard Deviation); unit: units on a scale] — The TRSI is a 24-item self-report measure assessing trauma-related shame on a 4-point Likert scale (Not true of me=0, Somewhat true of me=1, Mostly true of me=2, Completely true of me=3). A total shame score is summed ranging from 0-72 which higher scores reflecting a greater level of trauma-related shame.
  units on a scale | 26.84 (20.09)
Self-Compassion Scale (SCS) [Mean (Standard Deviation); unit: units on a scale] — The SCS is a 26-item self-report questionnaire that measures the cognitions and emotions associated with compassionate and uncompassionate responses to feelings of personal inadequacy and general life difficulties. Scores for negative items representing uncompassionate self-responding are reverse-coded to indicate their absence. Responses are given on a 5-point scale from "1-Almost Never" to "5-Almost Always." A total mean score is generated with higher scores corresponding to greater levels of self-compassion. Consider scores 1.0-2.49=low, between 2.5-3.5= moderate, and 3.51-5.0=high.
  units on a scale | 2.27 (.64)

OUTCOME MEASURES:

1. Primary Outcome: Self-Compassion Scale (SCS); Change From Baseline in Self-Compassion at Post-treatment
Description: The Self-Compassion Scale (SCS) is a 26-item self-report questionnaire that measures the cognitions and emotions associated with compassionate and uncompassionate responses to feelings of personal inadequacy and general life difficulties. Scores for negative items representing uncompassionate self-responding are reverse-coded to indicate their absence. Responses are given on a 5-point scale from "1-Almost Never" to "5-Almost Always." A total mean score is generated with higher scores corresponding to higher levels of self-compassion. Consider scores 1.0-2.49 to be low, between 2.5-3.5 to be moderate, and 3.51-5.0 to be high.
Time Frame: Post-Tx (8-10 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement (SEM) for the total self-compassion score on the SCS. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to post-treatment was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MSC)
Number analyzed (Participants) | 14
score on a scale | 0.45 (0.21)

2. Primary Outcome: Self-Compassion Scale (SCS); Change From Baseline in Self-Compassion at 1 Month Follow-up
Description: as for outcome 1
Time Frame: 1-Month Follow-up (12-14 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement for the total self-compassion score on the SCS. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to one-month follow-up was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Groups:
- Mindful Self-Compassion Intervention: Mindful Self-Compassion: Mindful Self-Compassion Intervention
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | 1.26 (0.21)

3. Primary Outcome: Trauma-Related Guilt Inventory (TRGI) - Distress Scale; Change From Baseline in Trauma-related Guilt Distress at Post-treatment
Description: The TRGI distress subscale is made up of 6 items (e.g., "I experience severe emotional distress when I think about what happened"). Respondents rate each statement using a 5-point Likert scale to indicate the degree to which they believe the statement is true about themselves (i.e., Extremely True=4, Very True=3, Somewhat True=2, Slightly True=1, or Never True=0). The items are summed and divided by 6 to create an average score raging from 0-4 with higher scores reflecting higher levels of distress.
Time Frame: Post-Tx (8-10 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement for the Distress subscale on the TRGI. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to post-treatment was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion (MSC)
Number analyzed (Participants) | 14
score on a scale | -0.28 (0.34)

4. Primary Outcome: Trauma-Related Guilt Inventory (TRGI) - Distress Scale; Change From Baseline in Trauma-related Guilt at 1-Month Follow-up
Description: as for outcome 3
Time Frame: 1-Month Follow-up (12-14 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement for the Distress subscale on the TRGI. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to 1-month follow-up was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | -0.45 (0.34)

5. Primary Outcome: Trauma-Related Shame Inventory (TRSI); Change From Baseline in Trauma-related Shame at Post-treatment Follow-up
Description: The TRSI is a 24-item self-report measure assessing trauma-related shame on a 4-point Likert scale (Not true of me=0, Somewhat true of me=1, Mostly true of me=2, Completely true of me=3). A total shame score is summed ranging from 0-72 which higher scores reflecting a greater level of trauma-related shame.
Time Frame: Post-Tx (8-10 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement for the TRSI sum score. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to post-treatment was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | -5.94 (3.04)

6. Primary Outcome: Trauma Related Shame Inventory (TRSI); Change From Baseline in Trauma-related Shame at 1-Month Follow-up
Description: as for outcome 5
Time Frame: 1-Month Follow-up (12-14 weeks post baseline)
Population: The investigators examined clinically meaningful change among treatment completers with complete pre- and post-treatment data using the standard error of measurement for the TRSI sum score. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to one-month follow-up was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | -8.46 (3.04)

7. Secondary Outcome: Clinician Administered PTSD Scale for Diagnostic and Statistical Manual-5 (DSM-5); Change From Baseline in PTSD Symptoms at Post-Treatment
Description: The Clinician Administered PTSD Scale for DSM-5 (CAPS-5) is a semi-structured interview used to assess PTSD diagnostic criteria and severity. The CAPS assesses each of the 20 items from the DSM-5 criteria B, C, D, and E. The assessor combines information about frequency and intensity of an item into a single severity rating (0=Absent; 1=Mild/subthreshold; 2=Moderate/threshold; 3=Severe/markedly elevated; 4=Extreme/incapacitating). CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms (range = 0-80). Similarly, CAPS-5 symptom cluster severity scores are calculated by summing the individual item severity scores for symptoms corresponding to a given DSM-5 cluster: Criterion B (items 1-5); Criterion C (items 6-7); Criterion D (items 8-14); and, Criterion E (items 15-20). Higher scores indicate worse PTSD symptoms.
Time Frame: Post-Tx (8-10 weeks post baseline)
Population: Clinically meaningful change among treatment completers with complete pre- and post-treatment data was examined using the standard error of measurement for the CAPS total severity sum score. The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to post-treatment for the CAPS total severity sum score was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | -5.86 (4.28)

8. Secondary Outcome: Clinician Administered PTSD Scale (CAPS-5); Change From Baseline in PTSD Symptoms at 1-Month Follow-up
Description: as for outcome 7
Time Frame: 1-Month Follow-up (12-14 weeks post baseline)
Population: Clinically meaningful change among treatment completers with complete pre- and post-treatment data was examined using the standard error of measurement for the CAPS total severity sum score. We defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to one-month post-treatment for the CAPS total severity sum score was calculated.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
score on a scale | -8.96 (4.28)

9. Secondary Outcome: Timeline Follow-back; Change From Baseline in Days Used Alcohol (Past 90 Days) at Post-treatment
Description: The Timeline Follow-back (TLFB) is a drinking assessment method that obtains estimates of daily drinking. The TLFB evaluates alcohol and other substance use during the previous 90 days. Using a calendar, people provide retrospective estimates of their daily drinking over a specified time period. The TLFB was used to establish: days respondents used alcohol.
Time Frame: Post-Tx (8-10 weeks)
Population: Clinically meaningful change among treatment completers with complete pre- and post-treatment data was examined using the standard error of measurement for days used alcohol (last 90 days; TLFB). The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to post-treatment for the days used alcohol was calculated.
Measure: Mean (Standard Error); unit: days used alcohol
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
days used alcohol | -24.30 (15.8)

10. Secondary Outcome: Timeline Follow-Back (TLFB); Change From Baseline in Days Used Alcohol (Past 90 Days) at 1 Month Follow Up
Description: The Timeline Follow-back (TLFB) is a drinking assessment method that obtains estimates of daily drinking. The TLFB evaluates alcohol and other substance use during the previous 90 days. Using a calendar, people provide retrospective estimates of their daily drinking over a specified time period. The TLFB was used to establish: number of days respondents used alcohol.
Time Frame: 1-Month Follow-up (12-14 weeks post baseline)
Population: Clinically meaningful change among treatment completers with complete pre- and post-treatment data was examined using the standard error of measurement for days used alcohol (last 90 days; TLFB). The investigators defined meaningful change as a reduction in scores by at least one SEM. The mean difference from baseline to one-month follow-up for the days used alcohol was calculated.
Measure: Mean (Standard Error); unit: days used alcohol
Arm/Group | Mindful Self-Compassion Intervention
Number analyzed (Participants) | 14
days used alcohol | -26.20 (15.8)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from participant enrollment (baseline) through one-month follow-up (approximately 12-14 weeks).
Arm/Group | Mindful Self-Compassion (MSC)
All-Cause Mortality (participants affected / at risk) | 2/26
Serious Adverse Events (participants affected / at risk) | 1/26
Other Adverse Events (participants affected / at risk) | 1/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Self-Compassion (MSC) (N=26)
Hospitalization/Medical (General disorders) | 1 (1) — Veteran was hospitalized at VA Medical Center after complaints of syncope to monitor heart rhythms and vitals.The Institutional Review Board (IRB) determined that this event was unrelated to the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindful Self-Compassion (MSC) (N=26)
Incarceration (Psychiatric disorders) | 1 (1) — Veteran incarcerated; event was not serious, unexpected, and deemed unlikely to be related to the study by the IRB. No changes to the study protocol or consent were required.

LIMITATIONS AND CAVEATS:
1) Sample size was small and consisted solely of male veterans. Future research should include more diverse samples to examine cultural and gender differences in treatment engagement and tolerability of MSC. 2) The current study lacks the experimental rigor associated with a randomized controlled trial. Findings regarding clinically meaningful change should be viewed as preliminary and in need of further study within the context of a larger efficacy trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT03681288/Prot_SAP_000.pdf